CLINICAL TRIAL: NCT04538170
Title: Neuropathic Pain After Orchidectomy and Sex Reassignment Surgery
Acronym: NPASRS
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 611/2013BO2
Record Dates: First submitted 2019-08-09; First posted 2020-09-04 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2014-08

CONDITIONS: Neuropathic Pain; Phantom Pain; Sex Reassignment Surgery
MeSH Terms: conditions — Neuralgia; Phantom Limb

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ORC: Group orchidectomy following cancer
  Interventions: Behavioral: pain after surgery
- GAC: Group sex reassignment surgery
  Interventions: Behavioral: pain after surgery

INTERVENTIONS:
Behavioral: pain after surgery

SUMMARY:
Phantom pain is associated with cortical reorganization after amputation. This phenomenon should not play a role in transsexual women, since the cortical representation of the male sex organs is presumably altered. The study investigates the incidence of phantom pain in this patient population.

For this study the following question should be investigated:

Is the incidence of phantom pain and local chronic postsurgical pain lower in sex reassignment surgery from male to female compared to inguinal tumor orchidectomy?

DETAILED DESCRIPTION:
Phantom pain is a common and much studied phenomenon after amputation.The loss of visceral organs is also associated with phantom pain. Under entirely different conditions than the removal of a tumorous testicle, sex reassignment surgery from male to female sex occurs in transsexual women. In this operation, parts of the penis and both testicles are removed and a plastic surgical transformation is made into a female genital.The surgical trauma is greater compared to an orchidectomy.

The sex reassignment surgery is expressly desired, the amputated tissues are rejected or perceived as not belonging to the patient's own body and thus do not appear as a loss. The group of patients with tumor orchidectomy acts as a control group.

In addition to the incidence of phantom pain and chronic local postoperative pain in comparison between the two groups, the secondary objectives of the study were defined as the occurrence of phantom pain, the type of pain and the intensity of pain.

Two patient groups were compared, the group after sex reassignment surgery (GAC) and the group after inguinal orchidectomy for testicular tumor (ORC).

A total of 265 transgender women were written to, 46 of whom had undergone surgery in Tübingen and 219 in Munich. The operations took place between 2002 and 2014.

For the group of patients after orchidectomy, 158 men who had undergone surgery in Tuebingen between 2010 and 2014 were contacted by letter.

The pseudonymization was done with a combination of letters and numbers, which were created with a key generator program.

The patients received a questionnaire divided into several categories, these categories were questions on demography, pre- and postoperative pain as well as phantom pain, pain processing, quality of life, sex life and urological questions.

ELIGIBILITY:
Inclusion Criteria:

* Surgery at least 6 month before data collection
* german speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after surgery (orcidectomy and sex resignment surgery in the universtiy hospital of Tuebingen Department of Urology and the Hospital of Munich Bogenhausen Department of Urology
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Tuebingen, clinic of anästhesiology and intensiv care, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- (ORC) Orchiectomy Following Cancer: 158 men who had undergone tumor orchidectomy between 2010 and 2014
- (GAC) Group Sex Reassignment Surgery: 265 transsexual women who had undergone surgery between 2002 and 2014
Period: Overall Study
Arm/Group | (ORC) Orchiectomy Following Cancer | (GAC) Group Sex Reassignment Surgery
Started | 158 | 265
Completed | 54 | 55
Not Completed | 104 | 210
Not completed — Withdrawal by Subject | 104 | 210

BASELINE CHARACTERISTICS:
Groups:
- ORC Group Orchidectomy Following Cancer: Group orchidectomy following cancer
  pain after surgery
- GAC Group Sex Reassignment Surgery: Group sex reassignment surgery
  pain after surgery
- Total: Total of all reporting groups
Arm/Group | ORC Group Orchidectomy Following Cancer | GAC Group Sex Reassignment Surgery | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.7) | 48.8 (10.1) | 46.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 55 | 109
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Phantom Pain
Description: Number of patients with phantom pain of testis
Time Frame: a minimum of 6 month post-surgery up to 5 years postsurgery
Measure: Count of Participants; unit: Participants
Groups:
- ORC Group Orchidectomy Following Cancer: phantom pain of testis after surgically removal
- GAC Group Sex Reassignment Surgery: pantom pain of testes after surgically removal
Arm/Group | ORC Group Orchidectomy Following Cancer | GAC Group Sex Reassignment Surgery
Number analyzed (Participants) | 54 | 55
Participants | 6 | 0
Statistical Analysis 1: Comparison: ORC Group Orchidectomy Following Cancer vs GAC Group Sex Reassignment Surgery; Preliminary work showed that approximately 25% of patients report phantom pain after orchidectomy. A difference of 20% between the GAC and ORC groups was considered relevant. Power was set to 80% and the significance level to 5%, resulting in a minimum of 40 women to be recruited, which was fulfilled; Test type: Superiority; p = 0.013, Fisher Exact — threshold for statistical significance

2. Secondary Outcome: Functional Outcome
Description: Number of Participants with Incontinence, Difficult Urination, Stenosis of Urethra, Spraying of Urine and/or Corrective Surgery"
Time Frame: a minimum of 6 month post-surgery up to 5 years postsurgery
Measure: Count of Participants; unit: Participants
Groups:
- ORC Group Orchidectomy Following Cancer; GAC Group Sex Reassignment Surgery: patients should give information about any type of incontinence
Arm/Group | ORC Group Orchidectomy Following Cancer | GAC Group Sex Reassignment Surgery
Number analyzed (Participants) | 54 | 55
Participants
  Incontinence | 1 | 7
  difficult urination | 2 | 5
  stenosis of the urethra | 0 | 11
  spraying of urine | 0 | 11
  corrective surgery | 3 | 19

3. Secondary Outcome: Incidence of Chronic Postoperative Pain
Description: Number of patients with chronic pain after surgery and differences between the two groups
Time Frame: a minimum of 6 month post-surgery up to 5 years postsurgery
Measure: Count of Participants; unit: Participants
Groups:
- ORC Group Orchidectomy Following Cancer; GAC Group Sex Reassignment Surgery: chronic pain in the region of surgery but not phantom pain
Arm/Group | ORC Group Orchidectomy Following Cancer | GAC Group Sex Reassignment Surgery
Number analyzed (Participants) | 54 | 55
Participants | 13 | 15

ADVERSE EVENTS:
Time Frame: a minimum of 6 month post-surgery up to 5 years postsurgery
Groups:
- GAC Gender Reassignment Surgery: 55 transsexual women who had undergone gender reassignment surgery answer a questionnaire
- ORC Patients After Inguinal Orchidectomy for Testicular Tumor: 54 patients after inguinal orchidectomy for testicular tumor, answer a questionnaire
Arm/Group | GAC Gender Reassignment Surgery | ORC Patients After Inguinal Orchidectomy for Testicular Tumor
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

LIMITATIONS AND CAVEATS:
The response rate could influence the result. One reason could be the large period of time between the operation and data collection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT04538170/Prot_SAP_000.pdf